CLINICAL TRIAL: NCT04059471
Title: Non- Inferiority Fractional-doses Trial for Yellow Fever Vaccine
Acronym: NIFTY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: KEMRI-Wellcome Trust Collaborative Research Program (Other); Institut Pasteur (Industry); MRC/UVRI and LSHTM Uganda Research Unit (Other); Epicentre, Paris, France. (Unknown)
Responsible Party: Principal Investigator, George Warimwe, PhD, Professor, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OxTREC Ref: 2-19; SERU 3797 (Other: KEMRI, Kenya); HS 2596 (Other: UNCST, Uganda); MUREC 1/7 (Other: MUST-REC, Uganda); ECCT/19/03/04 (Other: Pharmacy and Poisons Board, Kenya)
Record Dates: First submitted 2019-07-26; First posted 2019-08-16 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Yellow Fever
Keywords: Yellow Fever vaccine; Fractional doses; Yellow Fever; Vaccine dose
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Intervention Model Description: Adult participants (n=480) will be randomized for vaccination with full standard dose or with 1000, 500 or 250 IU (i.e. 4 arms) with a 1:1:1:1 allocation ratio. Results for the safety and primary outcome of the adult study will then be reviewed by the DSMB, and the lowest non-inferior dose in the adult study selected for assessment in children aged 9 months to 5 years (n=420) in comparison to full standard dose (i.e. 2 arms) with a 1:1 allocation ratio.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and participants will be blinded to the allocations. Only the pharmacist and the nurse administering the vaccine will be unblinded. The allocation will be to one of the four treatment arms per a computer-generated randomization schedule. Allocations will be concealed until a member of the unblinded study team scratches the randomization booklet to reveal the participants' randomization arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Dose (Active Comparator): Yellow fever vaccine, Institut Pasteur, standard dose as release by manufacturer will be administered subcutaneously once.
  Interventions: Biological: Yellow fever vaccine, Institut Pasteur
- Fractional dose (1000 IU/dose) (Experimental): Yellow fever vaccine, Institut Pasteur, will be titrated to about 1000IU/dose and administered subcutaneously once.
  Interventions: Biological: Yellow fever vaccine, Institut Pasteur
- Fractional dose (500 IU/dose) (Experimental): Yellow fever vaccine, Institut Pasteur, will be titrated to about 500IU/dose and administered once.
  Interventions: Biological: Yellow fever vaccine, Institut Pasteur
- Fractional dose (250 IU/dose) (Experimental): Yellow fever vaccine, Institut Pasteur, will be titrated to about 250IU/dose and administered once.
  Interventions: Biological: Yellow fever vaccine, Institut Pasteur

INTERVENTIONS:
Biological: Yellow fever vaccine, Institut Pasteur — Full dose and 500IU/dose
  Other Names: Children sub-study

SUMMARY:
In the recent past there has been a number of large urban Yellow Fever outbreaks in sub-Saharan Africa, tropical South Americas, The demand for Yellow Fever vaccines in response to the large urban outbreaks occurring concurrently and the risk of further spread through Africa and to Asia was larger than the available global supply. In this situation, the World Health Organisation (WHO) developed recommendations for the use of fractional doses of Yellow Fever vaccine as a dose-sparing strategy. These recommendations were based on data from a limited number of clinical trials, none of which had been conducted in Africa. This was due to the uncertainties on the minimum dose requirement.

Our study complements a study which is comparing full standard dose to 1/5th of standard dose of all four WHO-prequalified YF vaccines in adults (ClinicalTrials.gov number: NCT02991495), and is currently ongoing at KEMRI CGMRC and Epicentre, Mbarara which is designed to answer questions on the use of current stock of YF vaccines with a potency as close as possible to each manufacturers' minimum release. Data from this trial will inform a WHO recommendation on using 1/5th of the current standard dose of vaccine for outbreak control. However, since many vials will contain excess YF vaccine such that 1/5th of a vial is likely to be substantially above the current minimum potency requirements, these data may not be scientifically explanatory regarding the minimum dose required for preventive use.

The new complementary study, aims to determine the lowest YF vaccine dose that is non-inferior to the current standard full dose among populations in sub-Saharan Africa. The study will be conducted in Kenya (KEMRI Center for Geographical Medicine Research-Coast (CGMR-C), Kilifi) and Uganda (Epicentre, Mbarara) with trial participants recruited at both sites, using vaccine from one WHO-prequalified manufacturer (Institut Pasteur de Dakar, Senegal (IPD)).

DETAILED DESCRIPTION:
Yellow fever (YF) is a disease caused by a mosquito-borne flavivirus that is endemic in sub-Saharan Africa and tropical South America. Ninety percent of YF cases are in Africa where YF virus is transmitted by different mosquito genera in three recognized transmission cycles. A sylvatic cycle involves transmission between forest-dwelling mosquitoes (Haemagogus spp) and non-human primate reservoirs, with sporadic incidental transmission to humans (e.g. forest workers). An intermediate cycle, occurring only in Africa, involves mosquito transmission between non-human primates and humans, or human-to-human transmission among humans living or working close to forested areas. An urban cycle involves transmission between humans and urban mosquito vectors, primarily Aedes aegypti, and occurs when a viraemic person, infected in the sylvatic or intermediate cycle, introduces YF virus to areas with a large non-immune population and A. aegypti vectors resulting in disease outbreaks.

Infection with YF virus is characterised by a wide range of manifestations, ranging from subclinical infection with mild and non-specific symptoms, to severe, life-threatening illness with jaundice, renal failure and haemorrhage.

A highly effective vaccine is available for use against YF in adults and children aged ≥9 months. The vaccine is a freeze-dried preparation of live attenuated YF virus strain 17D, which was developed in 1937 and is produced by four WHO-prequalified manufacturers. A single dose of YF vaccine is considered sufficient to confer life-long protective immunity against all seven known genotypes of wild-type YF virus. Protective levels of YF virus neutralizing antibodies are developed in 80-100% vaccine recipients within 10 days after vaccination, and in 99% within a month.

Although fractional dosing has recently been used in vaccination campaigns in Kinshasa and Brazil in 2016, 2017 and 2018, WHO recommendations were based on a limited number of clinical studies and important data gaps remain.

fractional vaccine dosing is compounded by the uncertainty surrounding minimum dose requirements.

This study therefore aims to determine the lowest dose in International Units (IU/dose) that is non-inferior to the standard full dose among populations in sub-Saharan Africa. The data generated in this study will provide information regarding the re-definition of the minimal dose and potency requirements of the vaccine. The study will also provide further confidence in the use of fractional doses of YF vaccine during epidemics. In addition, the investigators will assess the range of views and perceptions of key stakeholders in vaccine policy and implementation on reduced vaccine dose usage during YF epidemics and for routine use.

. The study will be conducted at the KEMRI CGMRC in Kilifi, Kenya and at Epicentre in Mbarara, Uganda. Both these sites are already working together in an ongoing study (ClinicalTrials.gov number: NCT02991495).

Adult participants (n=480) will be randomized for vaccination with full standard dose or with 1000, 500 or 250 IU (i.e. 4 arms) with a 1:1:1:1 allocation ratio. Results for the safety and primary outcome of the adult study will then be reviewed by the DSMB, and the lowest non-inferior dose in the adult study selected for assessment in children aged 9 months to 5 years (n=420) in comparison to full standard dose (i.e. 2 arms) with a 1:1 allocation ratio. The determination of the non-inferior dose to use in children will be made by the sponsor in discussion with the study Data Safety and Monitoring Board (DSMB), vaccine manufacturer and relevant stakeholders, and the final decision communicated to the various regulatory authorities as a notification (i.e. Scientific and Ethics Review Board (SERU) at KEMRI, Oxford Tropical Research Ethics Committee (OxTREC) and Pharmacy and Poisons board (PPB) for the Kilifi site, Mbarara University of Science and Technology's Research Ethics Committee (MUST-REC), Uganda National Council of Science and Technology (UNCST) and National Drug Authority (NDA) for the Mbarara site).

Adult vaccinees will be followed up for 2 years, and children for 1 year. There will be no gradual age de-escalation on the basis that there are few safety concerns with the full dose of YF vaccines, having been used in millions of children worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged ≥18 - <60 years of age.
* Children aged between 9 months and 12 months.
* HIV negative on serological screening OR HIV positive adults and children aged > 18 months on serological testing, and no symptoms suggestive of current clinical immunosuppression and cluster of differentiation-4 (CD4) count>200 (for adults) and CD4% > 25% (for children aged 9-12 months) within the last 6 months.
* Ability to provide informed consent to participate in the study

Exclusion Criteria:

* Known contraindications to YF vaccination such as allergies to egg protein and chicken products or any component of the vaccine (including gelatin, eggs, eggs products or chicken products), immunodeficiency, known thymus disorder, such as thymoma and myasthenia gravis
* Using corticosteroids or other immunosuppressive therapy
* Thymus disorder, such as thymoma and myasthenia gravis
* Acute febrile disease on the day of vaccination with temperature >37.5 degrees Celsius is a temporal contraindication.
* Previous YF vaccination
* Previous YF infection as determined from history
* Pregnancy (as determined by a urine test on the proposed day of vaccination) and lactating women
* Planning to migrate out of the study areas before the end of the study follow-up
* Planning to travel to a country requiring YF vaccination certificate within the first year after vaccination.
* Any condition or criteria, including acute or chronic clinically significant abnormality that in the opinion of the investigator might compromise the wellbeing of the volunteer or interfere with the outcome of the study.

Ages: 9 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 900 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2023-06-24 (Actual)

PRIMARY OUTCOMES:
The proportion of vaccinees that seroconverts as measured by Plaque Reduction Neutralisation Test (PRNT-50) | 28 days post vaccination
  PRNT-50 will be used to quantify functional antibodies by neutralisation of the virus

SECONDARY OUTCOMES:
Duration of immunity as measured by PRNT | 10 days, 28 days, 1 year and 2 years (adults)
  To describe the longevity of functional antibodies post-vaccination with the different doses as measured by PRNT
Change in the geometric mean fold of the antibody titre as measured by PRNT | Baseline and 28 days after vaccination
  To describe change in the geometric mean antibodies between baseline and 28 days after vaccination.
Other flavivirus antibodies interference as tested by neutralisation tests | Baseline and 28 days after vaccination
  To measure the impact of antibodies to other flaviviruses (including dengue, West Nile and zika viruses) on the baseline sample on YF vaccine immunogenicity 28 days after vaccination by pairwise comparison.
Post-vaccination viremia as measured by quantitative Polymerase Chain Reaction (PCR) | baseline, and on days 2, 3, 4, 5, 6, 7 and 10 after vaccination
  To assess post-vaccination control of viremia by different vaccine doses by sparse sampling
Changes in cellular immunology | baseline and days 10 and 28 post-vaccination.
  To determine the change in T and B cell immune responses between baseline and days post-vaccination
Changes in biomarkers | Baseline, and on days 2, 3, 4, 5, 6, 7,10 and 28 after vaccination
  To determine the change in serum biomarkers levels (including, TNF, INF-γ, IL-2, IL-4, IL-5, IL-10, IL-8/CXCL-8, MCP-1/CCL-2, MIG/CXCL-9 and IP-10/CXCL-10) between baseline and post-vaccination by pairwise comparison.
Safety of different doses as described by the occurrence of adverse events (AE) and serious adverse events. | 28 days after vaccination and an average of 1 year for the adult study and two years for the children study. .
  To assess the occurrence of adverse events (AE) over 28 days after vaccination and serious adverse events throughout the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bejon, PhD, Study Director — University of Oxford
Locations (2):
- KEMRI-Wellcome Trust Research Programme, Kilifi, Coast, Kenya
- Epicentre, Mbarara., Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will be de-identified and coded before sharing.

REFERENCES:
- [Derived] Kimathi D, Juan-Giner A, Bob NS, Orindi B, Namulwana ML, Diatta A, Cheruiyot S, Fall G, Dia M, Hamaluba MM, Nyehangane D, Karanja HK, Gitonga JN, Mugo D, Omuoyo DO, Hussein M, Oloo E, Kamau N, Wafula J, Bendera J, Silvester N, Mwavita J, Joshua M, Thuranira JM, Agababyona C, Ngetsa C, Aisha N, Moki F, Buluku T, Munene M, Mwanga-Amumpaire J, Lutwama J, Kayiwa J, Kamaara E, Barrett AD, Kaleebu P, Bejon P, Sall AA, Grais RF, Warimwe GM. Low-dose yellow fever vaccination in infants: a randomised, double-blind, non-inferiority trial. Lancet. 2026 Jan 13:S0140-6736(25)02069-0. doi: 10.1016/S0140-6736(25)02069-0. Online ahead of print. PMID 41544642
- [Derived] Kimathi D, Juan-Giner A, Bob NS, Orindi B, Namulwana ML, Diatta A, Cheruiyot S, Fall G, Dia M, Hamaluba MM, Nyehangane D, Karanja HK, Gitonga JN, Mugo D, Omuoyo DO, Hussein M, Oloo E, Kamau N, Wafula J, Bendera J, Silvester N, Mwavita J, Joshua M, Mwendwa J, Agababyona C, Ngetsa C, Aisha N, Moki F, Buluku T, Munene M, Mwanga-Amumpaire J, Lutwama J, Kayiwa J, Kamaara E, Barrett AD, Kaleebu P, Bejon P, Sall AA, Grais RF, Warimwe GM; NIFTY Investigators. Low-Dose Yellow Fever Vaccine in Adults in Africa. N Engl J Med. 2025 Feb 20;392(8):788-797. doi: 10.1056/NEJMoa2407293. PMID 39970397
- [Derived] Kimathi D, Juan A, Bejon P, Grais RF, Warimwe GM; YEFE and NIFTY vaccine trials teams. Randomized, double-blinded, controlled non-inferiority trials evaluating the immunogenicity and safety of fractional doses of Yellow Fever vaccines in Kenya and Uganda. Wellcome Open Res. 2019 Nov 20;4:182. doi: 10.12688/wellcomeopenres.15579.1. eCollection 2019. PMID 31984244